CLINICAL TRIAL: NCT03394820
Title: Determining the Optimal Time of IV Dexamethasone Administration for Prolongation of Peripheral Nerve Block
Brief Title: The Optimal Time of IV Dexamethasone Administration for Prolongation of Peripheral Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 16-5116-A
Record Dates: First submitted 2017-09-07; First posted 2018-01-09 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Nerve Block Prolongation; Hand Injury Wrist
Keywords: Dexamethasone; Supraclavicular block
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: the patients will be randomized into four differently times groups. The patients will receive dexamethasone either 1 hour before the block, during the block, 1 hour after the block or 2 hours after the block
Who Masked: Care Provider, Investigator
Masking Description: The patient will be randomized prior to surgery. The pre-randomized envelope will be given to the anesthesia assistant by the blinded research associate. The anesthesia assistant will then prepare the four mini-bags labelled with the time each bag should be hung.The four bags will include 1 active drug and 3 placebo, to administer to the patient. The clinical fellow who will be administering the four doses will be blinded, as well as the research associate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- dexamethasone 1 hour prior to block (Active Comparator): The patient will receive dexamethasone through IV one hour prior to receiving their block. During the patient's block, 1 hour after and 2 hours after the block the patient will receive infusions of normal saline to maintain the blind.
  Interventions: Drug: Dexamethasone
- dexamethasone during the block (Experimental): The patient will receive dexamethasone through IV at the same time the patient has the SCB done. One hour prior to the block, one hour after the block and 2 hours after the block the patient will receive infusions of normal saline to maintain the blind.
  Interventions: Drug: Dexamethasone
- dexamethasone 1 hour after block (Active Comparator): The patient will receive dexamethasone through IV one hour after the block has been administered. One hour prior to block, during the block and two hours after the block the patient will receive normal saline to maintain the blind.
  Interventions: Drug: Dexamethasone
- dexamethasone 2 hours after block (Active Comparator): The patient will receive dexamethasone 2 hours after the block has been administered. One hour prior to the block, during the block and one hour after the block the patient will receive normal saline to maintain the blind.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — The intervention is the time when dexamethasone is administered

SUMMARY:
The purpose of this study is to determine the optimal timing of IV dexamethasone for prolongation of ultrasound (US) guided supraclavicular brachial plexus block (SCB) in patients undergoing unilateral hand or forearm surgery at the Toronto Western Hospital. Investigators seek to answer which timing of IV dexamethasone will provide the maximum block prolongation. Investigators hypothesize that IV dexamethasone administered either before or after the block will further extend the duration of analgesia provided.

DETAILED DESCRIPTION:
This is a prospective double-blind randomized trial to evaluate the optimal timing of IV dexamethasone. All patients undergoing isolated hand or forearm surgery under anesthetic will be approached to participate. The patients will be consented on the day of surgery; all patients will be fully informed of the procedures involved in the study. Once the patient has consented to the study, they will be randomized to receive dexamethasone at one of four different times: 1 hour before the block, during the block, 1 hour after the block and 2 hours after the block.

In accordance with routine pre-block management, non-invasive blood pressure, electrocardiogram and pulse oximetry will be applied and intravenous access secured on the non-operative side for infusion of a 0.9% saline solution. Prior to block performance all patients will receive intravenous midazolam 1 - 4mg IV and / or fentanyl 25mcg IV for anxiolysis and analgesia, respectively, as needed. The US-guided SCB will be performed under sterile conditions by a staff regional anesthetist, regional anesthesia fellow or a directly supervised resident with experience of at least 10 US-guided SCB performed for each approach. Ultrasound examination above the clavicle will be performed using a high frequency linear probe (5 - 12 MHz range) with either a Philips, Sonosite or GE ultrasound machine. The brachial plexus, subclavian artery, first rib and pleura will be identified in the supraclavicular fossa. A 22 - gauge insulated 50mm needle (Stimuplex, Braun Medical, Bethlehem, PA) will be introduced in plane with the US and advanced to puncture the brachial plexus sheath. Typically this is accompanied by a palpable 'fascial click'. A small amount (0.5-1ml) of local anesthetic will be incrementally injected for needle tip hydro-location and/or hydro-dissection at the discretion of the operator. After placing the needle tip near the intersection of the first rib and the lateral aspect of the subclavian artery ('corner pocket') 30mls of 0.5% bupivacaine will be injected incrementally in 5ml aliquots with intermittent aspiration for blood.

A blinded research associate will evaluate sensory loss and motor blockade every 5 minutes until surgery starts.

Supplemental mask oxygen IV fluid replacement and full monitoring will be continued intraoperatively. Intravenous sedation will be used at the discretion of the attending anesthetist and according to the patient's wishes as is the standard of care at our institution. The dose of sedative and / or analgesic drugs will be recorded. Attendants will be asked to avoid any intraoperative steroid therapy. Surgical duration will be recorded for comparative analysis and exclusion of cases <30 or >180 minutes.

Following surgery, patients will be transferred to the post-operative care unit (PACU) or fast-tracked for discharge directly from the day case unit. The onset time of surgical pain (if applicable) and first analgesic request will be recorded. Once oral intake is established, patients will receive one of two analgesic preparations as needed; Tylenol#3® (acetaminophen 300mg/codeine 30mg/caffeine 15mg per tablet) or Percocet® (acetaminophen 325mg/oxycodone HCl 5mg) if intolerant to codeine. Patients will be evaluated at 1 and 2 hours postoperatively noting pain scores, analgesics received, block density and recovery criteria.

On discharge from hospital, patients will receive a prescription of Tylenol#3® as needed or Percocet® if intolerant to codeine. Patients will be given a home diary to complete. Patients will be requested to record the time at which they first experience pain at the surgical site, the time of first analgesic use and the time when they regain normal (or baseline equivalent) strength in their fingers. Patients will be asked to complete diary entries at 8 hrs, 24hrs, 48hrs and 7 days post operatively. They will be asked to document their visual analogue (VAS) pain score, cumulative analgesic consumption, side effects (numbness / tingling in the operative arm, weakness in the operative arm, pain around the injection site, bruising around the injection site, nausea and vomiting) and current VAS for satisfaction pertaining to the analgesia received. Patients will be telephoned at the aforementioned times to collect data from the diary, which was found the most reliable method of data collection during a previous study. Finally, patients will be phoned at 3 months to ensure no long - term numbness or weakness related to the nerve block.

The doses of oral codeine or oxycodone consumed by each patient will be converted into equi-analgesic doses of oral morphine sulphate in order to facilitate comparison between groups.

Sample size for the study:

A total of 220 participants will be randomized to receive dexamethasone at one of four different time points: 1 hour before the block, during the block, 1 hour after the block and 2 hours after the block.

ELIGIBILITY:
Inclusion Criteria:

* Patients having isolated hand or forearm surgery under anesthetic ultrasound - guided SCB
* ASA class I - III
* Age 18 - 80 years, inclusive
* BMI <35

Exclusion Criteria:

* Pre - existing neuropathy or neurological deficit in the distribution of the nerves to be anaesthetized
* Contra-indication to regional anesthesia / supraclavicular brachial plexus blockade; bleeding diathesis, coagulopathy, local infection, severe respiratory disease
* Anatomical deformity precluding block placement
* Patients with a known history of hypersensitivity to local anesthetics and / or dexamethasone
* Patients taking steroid therapy
* Positive pregnancy test
* Inability to give informed consent
* Anticipated surgical time < 30 or > 180 minutes
* Any known contraindication for IV dexamethasone as per the product monograph:bacteremia and systemic fungal infections, hypersensitivity to any of the products components, gastric and duodenal ulcers, certain viral infections (i.e. varicella & herpes genitalis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Block Duration | from time from the end of the local anesthetic injection to patient report full freezing gone
  Sensory block duration i.e., time from the end of the local anesthetic injection (US - guided SCB) to the onset of pain at the surgical site.

SECONDARY OUTCOMES:
Block onset time | from time from the end of the local anesthetic injection (US - guided SCB) to surgical procedure start
  motor and sensation will be tested after the block is administered
Measures of recovery | 1 hour after surgery
  total opioid consumption (total PO morphine equivalent post operative)
Measures of recovery | 1 hour after surgery
  pain scores (0 no pain to 10 worst pain possible)
Time of first analgesic consumption | end of surgery to one week after surgery
  time from block onset to first outpatient analgesic
Motor block duration | one week after surgery
  patient reported recovery of normal finger strength
Opioid consumption | time of block to 1 week after
  The amount of opioids the the patient consumes post-operatively will be monitored
VAS Pain scores | end of surgery to one week post- op
  subjective pain scores
Patient satisfaction | after surgery to one week after surgery
  Subjective reported satisfaction at specific time points
Frequency and severity of adverse symptoms | one week post operatively
  adverse symptoms related to the block
Pain Questionaire | Three months after surgery
  presence or absence of pain post-operatively
total opioid consumption | 1 hour after surgery
  total PO morphine equivalent post operative

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD,FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hopspital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grass A, Chan V, Short AJ, Busser MJ, Chin KJ, Chowdhury J, Huszti E, Li Q, Perlas A. Timing of intravenous dexamethasone and analgesia after brachial plexus block: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2024 Dec 25:rapm-2024-105923. doi: 10.1136/rapm-2024-105923. Online ahead of print. PMID 39721764